CLINICAL TRIAL: NCT04143841
Title: A Pilot Study to Evaluate the Safety and Effectiveness of the Viveye Ocular Magnetic Neurostimulation System (OMNS) for the Management of Severe Dry Eye Disease
Brief Title: Viveye Ocular Magnetic Neurostimulation System (OMNS) for the Management of Severe Dry Eye Disease
Acronym: OMNS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Financial constraints
Sponsor: Epitech Mag Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLP-10003
Record Dates: First submitted 2019-09-24; First posted 2019-10-29 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Dry Eye Syndromes; ATD; Sjogren's Syndrome
MeSH Terms: conditions — Dry Eye Syndromes; Sjogren's Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single treatment (Active Comparator): A single treatment will be administered for both eyes for each subject. The treatment will be administered for 11 minutes per treated eye.
  Interventions: Device: Viveye OMNS treatment
- Single sham treatment (Sham Comparator): A single treatment will be administered for both eyes for each subject. The treatment will be administered for 11 minutes per treated eye.
  Interventions: Device: Viveye OMNS sham treatment

INTERVENTIONS:
Device: Viveye OMNS treatment — The Viveye OMNS treatment ( ~30 min) will be applied once, during the treatment visit only
  Arms: Single treatment
Device: Viveye OMNS sham treatment — The Viveye OMNS sham treatment ( ~30 min) will be applied once, during the treatment visit only
  Arms: Single sham treatment

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of Viveye OMNS non-invasive treatment for management of the signs and symptoms of severe dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, 18-80 years old
2. Subjects with severe aqueous deficient dry eye disease (concomitant meibomian gland disease is permitted):

   1. SPEED questionnaire score ≥ 10 AND
   2. Fluorescein Corneal Staining Score (FCSS) ≥ 5 NEI score in at least in one eye AND
   3. Schirmer score ≤ 10 mm in at least one eye (at screening or treatment day pre-treatment)
3. No contact lens wear for at least seven days prior to the Screening Visit and willingness to forego contact lens wear for the duration of the study;
4. Literacy, able to speak English or Hebrew, and able to complete questionnaires independently;
5. Willing and able to sign the informed consent form and deemed capable of complying with the requirements of the study protocol (tests and follow-up visits).

Exclusion Criteria:

1. Significant anterior blepharitis including signs of Demodex eyelid infection;
2. If the subject is using prescription dry eye ophthalmic drug such as Restasis (Cyclosporine A 0.05% ophthalmic emulsion), Xiidra (Lifitegrast), Cequa (Cyclosporine 0.09% ophthalmic solution), and the medication has not been used regularly for the past 3 months prior to screening visit;
3. Change in eye lubricant type usage in the last 1 month prior enrollment. Use of any device to manage DED within 1 month of Screening Visit;
4. Punctal plugs are present at screening that were inserted in the last 30 days prior enrollment, or intracanalicular plug that were inserted in the last 6 months in any eyelid;
5. Corneal transplant in either or both eyes;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2021-01-06 (Actual); Study Completion 2021-01-06 (Actual)

PRIMARY OUTCOMES:
Best corrected visual acuity (BCVA) | 12 weeks
  Frequency of treatment related deterioration in BCVA
Intraocular Pressure (IOP) | 12 weeks
  IOP results will be summarized descriptively. 95% confidence intervals for the difference between treatment arms at each visit will be presented, assuming t-distribution.
Slit lamp biomicroscopy | 12 weeks
  The percent related to worsening in ocular pathological changes observed
Rate of device/treatment related adverse events | 12 weeks
  Rate of device/treatment related Incidence of Adverse events (AE) will be presented in tabular form by seriousness, severity and relation to treatment
Fluorescein corneal staining | 12 weeks
  Change from baseline in fluorescein corneal staining score (NEI Scale 0-15) per treatment arm and visit (lower scores mean a better outcome.)
Ocular discomfort questionnaires | 12 weeks
  Change from baseline in ocular discomfort questionnaires (Standard Patient Evaluation of Eye Dryness - SPEED) per treatment arm and visit. score from 0 to 28, higher scores mean a worse outcome. (Reduction in SUM score = improvement)

CONTACTS AND LOCATIONS:
Locations (3):
- Israel (3):
  - E.Wolfson MC, Holon
  - SZMC, Jerusalem
  - Sourasky Medical Center, Tel Aviv